CLINICAL TRIAL: NCT04677543
Title: A Randomized, Double-Blind, Placebo-Controlled, Active Comparator, Multicenter Study to Validate Patient-Reported Outcome Instruments in Adult Subjects With Newly Diagnosed Nontuberculous Mycobacterial (NTM) Lung Infection Caused by Mycobacterium Avium Complex (MAC)
Brief Title: Validation of Patient Reported Outcome Measures in Participants With Nontuberculous Mycobacterial Lung Infection Caused by Mycobacterium Avium Complex
Acronym: ARISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: INS-415; 2020-002545-42 (EudraCT Number)
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Mycobacterium Infections, Nontuberculous
Keywords: Nontuberculous Mycobacterial Lung Infection; Mycobacterium avium complex; Psychometric validation; Patient-reported outcome
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous; Mycobacterium avium-intracellulare Infection | interventions — Azithromycin; Ethambutol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALIS + Background Regimen (Azithromycin + Ethambutol) (Active Comparator): Participants will be administered 590 mg of ALIS (amikacin liposome inhalation suspension) once daily. Participants will also be administered the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily.
  Interventions: Drug: ALIS; Drug: Azithromycin; Drug: Ethambutol
- ELC + Background Regimen (Azithromycin + Ethambutol) (Placebo Comparator): Participants will be administered ELC (empty liposome control), a matching placebo to ALIS, once daily. Participants will also be administered the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily.
  Interventions: Drug: Azithromycin; Drug: Ethambutol; Drug: ELC

INTERVENTIONS:
Drug: ALIS — Inhalation via nebulization over approximately 6 to 15 minutes.
  Other Names: Amikacin liposome inhalation suspension; ARIKAYCE®
  Arms: ALIS + Background Regimen (Azithromycin + Ethambutol)
Drug: Azithromycin — Oral tablet
  Other Names: AZI
Drug: Ethambutol — Oral tablet
  Other Names: ETH
Drug: ELC — Inhalation via nebulization over approximately 6 to 15 minutes.
  Other Names: Empty liposome control
  Arms: ELC + Background Regimen (Azithromycin + Ethambutol)

SUMMARY:
The primary objective of this study is to generate evidence demonstrating the domain specification (via modern psychometric methods), reliability, validity, and responsiveness (within-subject meaningful change) of the Patient-Reported Outcome (PRO) endpoints.

DETAILED DESCRIPTION:
Participants will also complete the EXAcerbations of Chronic Pulmonary Disease Tool (EXACT), EXACT Respiratory Symptoms (EXACT-RS), St. George Respiratory Questionnaire (SGRQ), Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue), Patient Global Impression of Severity - Respiratory (PGIS-Respiratory), and Patient Global Impression of Severity - Fatigue (PGIS-Fatigue) at baseline and throughout the study as anchors for the validation of the QoL-B and PROMIS F-SF 7a.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age (19 years or older in South Korea)
* Current diagnosis of Mycobacterium avium Complex (MAC) lung infection
* Positive sputum culture for MAC within 6 months prior to screening
* A chest computed tomography (CT) scan, read locally, within 6 months prior to Screening to determine presence and size of pulmonary cavities. Participants who do not have a chest CT scan within 6 months prior to Screening will be required to obtain a chest CT scan, read locally, during Screening
* Willingness and ability to adhere to prescribed study treatment during the study
* Ability to produce (spontaneously or with induction) approximately 2 mL of sputum for mycobacteriology at Screening
* Women of child-bearing potential (WOCBP) (ie, fertile following menarche and until becoming post-menopausal unless permanently sterile) and fertile men (ie, all men after puberty unless permanently sterile by bilateral orchidectomy) agree to practice a highly effective method of birth control from Day 1 to at least 90 days after the last dose. Examples of such birth controls are:

  * true abstinence (refraining from heterosexual intercourse during the entire study),
  * copper intrauterine device (IUD),
  * hormonal methods (levonorgestrel-releasing intrauterine system, progestogen implant, combined oral contraceptive pill [combined with barrier method]),
  * exclusive homosexual relationship, or
  * sole male partner who has undergone surgical sterilization with confirmation of azoospermia at least 3 months post procedure while participating in the study
* Provide signed informed consent prior to administration of study drugs or performing any study related procedure
* Be able to comply with study drugs use, study visits, and study procedures as defined by the protocol
* Men with partners who are WOCBP (pregnant or non-pregnant) agree to use condoms and non-pregnant partners should practice a highly effective method of birth control

Exclusion Criteria:

* Diagnosis of cystic fibrosis (CF)
* History of more than 3 MAC lung infections
* Received any mycobacterial antibiotic treatment for current MAC lung infection
* Refractory MAC lung infection, defined as having positive MAC cultures while being treated with a multidrug mycobacterial antibiotic treatment regimen for a minimum of 6 consecutive months and no documented successful treatment, defined as negative sputum culture for MAC and cessation of treatment
* Relapse of prior MAC lung infection, defined as positive sputum culture for MAC ≤ 6 months of cessation of prior successful treatment
* Evidence of any pulmonary cavity ≥ 2 cm in diameter, as determined by chest CT scan, read locally, within 6 months prior to Screening
* Radiographic finding of new lobar consolidation, atelectasis, significant pleural effusion, or pneumothorax during routine clinical care within 2 months prior to Screening
* Active pulmonary malignancy (primary or metastatic) or any malignancy requiring chemotherapy or radiation therapy within 1 year prior to Screening or anticipated during the study
* Acute pulmonary exacerbation (eg, chronic obstructive pulmonary disease [COPD] or bronchiectasis) requiring treatment with antibiotics, or corticosteroids (intravenous [IV] or oral), within 4 weeks prior to and during Screening
* Current smoker
* History of lung transplantation
* Prior exposure to amikacin liposome inhalation suspension (ALIS) (including clinical study)
* Known hypersensitivity or contraindications to use to ALIS, aminoglycosides, or any of their excipients
* Disseminated MAC infection
* Positive pregnancy test or lactation at Screening. All WOCBP will be tested. Women not of childbearing potential are defined as postmenopausal (ie, amenorrheic for 12 months without an alternative medical cause or confirmed by more than one follicle stimulating hormone [FSH] measurement), or naturally or surgically sterile through bilateral oophorectomy, hysterectomy, or bilateral salpingectomy. For women under the age of 45 years, confirmatory testing with FSH should be considered
* Administration of any investigational drug within 8 weeks prior to Screening
* Known or suspected acquired immunodeficiency syndromes (HIV-positive, regardless of CD4 counts). Other immunodeficiency syndromes that may interfere with study participation in the opinion of the Investigator.
* Current alcohol, medication, or illicit drug abuse
* Known and active COVID-19 infection
* MAC isolate with MIC for clarithromycin ≥ 32 µg/mL at Screening
* Known hypersensitivity or contraindications to use to ethambutol, azithromycin (including other macrolides or ketolides), or any of their excipients per local labeling guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (27):
  - USA008, Birmingham, Alabama
  - USA062, Fresno, California
  - USA048, San Diego, California
  - USA050, Stanford, California
  - USA023, Washington D.C., District of Columbia
  - USA003, Clearwater, Florida
  - USA072, Jacksonville, Florida
  - USA042, Kissimmee, Florida
  - USA039, Naples, Florida
  - USA014, St. Petersburg, Florida
  - USA067, Tampa, Florida
  - USA066, Augusta, Georgia
  - USA029, Rincon, Georgia
  - USA037, Kansas City, Kansas
  - USA017, Baltimore, Maryland
  - USA061, St Louis, Missouri
  - USA069, Hillsborough, New Jersey
  - USA065, Bayside, New York
  - USA011, New York, New York
  - USA051, Durham, North Carolina
  - USA025, Portland, Oregon
  - USA040, Philadelphia, Pennsylvania
  - USA044, Anderson, South Carolina
  - USA024, Charleston, South Carolina
  - USA022, Franklin, Tennessee
  - USA021, McKinney, Texas
  - USA052, Tyler, Texas
- ARG003, Córdoba, Argentina
- Australia (3):
  - AUS010, Chermside, Queensland
  - AUS011, Woolloongabba, Queensland
  - AUS008, Adelaide, South Australia
- AUT001, Linz, Austria
- Denmark (3):
  - DNK001, Roskilde, Zeeland
  - DNK004, Aalborg
  - DNK002, Aarhus
- Germany (5):
  - GER005, München, Bavaria
  - GER010, Immenhausen, Hesse
  - GER007, Hanover, Lower Saxony
  - GER011, Cologne, North Rhine-Westphalia
  - GER006, Dresden
- Israel (4):
  - ISR001, Ashkelon
  - ISR007, Haifa
  - ISR003, Petah Tikva
  - ISR004, Ramat Gan
- Italy (4):
  - ITA006, Modena, Emilia-Romagna
  - ITA005, Rome, Lazio
  - ITA008, Siena, Tuscany
  - ITA002, Milan
- New Zealand (3):
  - NZL003, Hastings, Hawkes's Bay
  - NZL002, Hamilton, Waikato Region
  - NZL001, Christchurch
- South Korea (3):
  - KOR005, Seongnam
  - KOR002, Seoul
  - KOR003, Seoul
- Spain (5):
  - ESP002, Barcelona
  - ESP003, Barcelona
  - ESP005, Girona
  - ESP001, Madrid
  - ESP004, Madrid
- Taiwan (3):
  - TWN004, Chiayi City, Chiayi
  - TWN005, Kaohsiung City
  - TWN002, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daley CL, Chalmers JD, Flume PA, Griffith DE, Hasegawa N, Morimoto K, Winthrop KL, Sheu CC, Avsar K, Andrisani D, Codecasa LR, Yuen DW, Hassan M, Nevoret ML, Mange K. Trial Conduct, Baseline Characteristics, and Symptom Burden of Patients in the ARISE Study. Pulm Ther. 2025 Jun;11(2):269-283. doi: 10.1007/s41030-025-00293-3. Epub 2025 Apr 8. PMID 40198465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this multi-centre study at different investigative sites from 22 December 2020 to 09 May 2023
Groups:
- ALIS + Background Regimen (Azithromycin + Ethambutol): Participants received 590 mg of amikacin liposome inhalation suspension (ALIS) once daily. Participants also received the background regimen of azithromycin 250 mg and ethambutol 15 milligrams per kilogram (mg/kg) tablets orally, once daily.
- ELC + Background Regimen (Azithromycin + Ethambutol): Participants received empty liposome control (ELC), a matching placebo to ALIS, once daily. Participants also received the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily.
Period: Overall Study
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Started | 48 | 51
Completed | 44 | 48
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Analysis Set comprises all participants who were randomized.
Groups:
- ALIS + Background Regimen (Azithromycin + Ethambutol): Participants received 590 mg of ALIS once daily. Participants also received the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily.
- ELC + Background Regimen (Azithromycin + Ethambutol): Participants received ELC, a matching placebo to ALIS, once daily. Participants also received the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily.
- Total: Total of all reporting groups
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol) | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (9.51) | 65.9 (12.27) | 67.4 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 45 | 77
  Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 45 | 48 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 12 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 41 | 39 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Psychometric Cross-Sectional Validation of Patient Reported Outcome (PRO): Patient Global Impression of Severity (PGI-S) Respiratory Scale Score at Baseline
Description: The PGI-S respiratory symptom is a self-reported scale to measure the severity of illness based on symptoms using a 5-point scale ranging from 1 to 5, (1=not at all, 2=mild, 3=moderate, 4=very severe, 5=extremely severe). Considering different aspects of breathing symptoms like congestion, cough, mucus, wheezing, shortness of breath, participants rated their symptom severity on the PGI-S respiratory symptom scale. Higher scores indicate greater symptom severity.
Time Frame: Baseline
Population: ITT Analysis Set comprises all participants who were randomized.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
score on scale | 2.5 (0.82) | 2.4 (0.90)

2. Primary Outcome: Psychometric Cross-Sectional Validation of PRO: PGI-S Fatigue Scale Score at Baseline
Description: The PGI-S fatigue is a self-reported scale to measure the severity of illness based on symptoms using a 5-point scale ranging from 1 to 5, (1=not at all, 2=mild, 3=moderate, 4=very severe, 5=extremely severe). Participants rated the severity of their fatigue on the PGI-S fatigue scale. Higher scores indicate greater fatigue severity.
Time Frame: Baseline
Population: ITT Analysis Set comprises all participants who were randomized.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- ALIS + Background Regimen (Azithromycin + Ethambutol): Participants received 590 mg of amikacin liposome inhalation suspension (ALIS) once daily. Participants also received the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily.
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
score on scale | 2.5 (0.99) | 2.5 (0.81)

3. Primary Outcome: Psychometric Cross-Sectional Validation of PRO: Quality of Life Questionnaire - Bronchiectasis (QoL-B) Respiratory Symptoms Scale Score at Baseline
Description: The QOL-B is a self-administered, PRO questionnaire used to assess symptoms, functioning, and health related quality of life in adults with lung conditions. The respiratory symptom domain of the QOL-B contains 9 items describing patient's self-assessment of her/his respiratory symptoms that affect daily life. For each of the 8 items (chest congestion, coughing, cough up mucus, shortness of breath with greater activity, wheezing, chest pain, shortness of breath when talking, woken up during night due to cough), scores ranged from 1 to 4 (1= lot, 2= moderate, 3= little, 4= not at all) and the sputum item based on the color ranged from 0=don't know,1=green with traces of blood/brownish dark,2=yellowish-green,3=clear to yellow,4=clear. The item scores were summed and then standardized on a 0 to 100-point scale to derive the domain score with higher scores representing fewer symptoms or better functioning and quality of life.
Time Frame: Baseline
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
score on scale | 63.04 (14.824) | 66.90 (15.673)

4. Primary Outcome: Psychometric Cross-Sectional Validation of PRO: Patient-Reported Outcome Measurement Information System - Fatigue-Short Form 7a (PROMIS F-SF 7a) Score at Baseline
Description: The PROMIS F-SF 7a is a self-administered questionnaire assessing a range of self-reported symptoms over the past 7 days, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities over 7 items. Response options are on a 5-point Likert scale, ranging from 1=never to 5=always. Total scores range from 7 to 35 and low scores represent less fatigue interference i.e., better symptoms.
Time Frame: Baseline
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
score on scale | 18.3 (5.76) | 18.6 (4.76)

5. Primary Outcome: Assessment of Test-Retest Reliability (TRTR) Reported as the Intraclass Co-relation (ICC) Estimate Among Participants Reporting no Change on Respiratory PGI-S Score Applied to QOL-B Respiratory Domain Score Between Screening and Baseline
Description: TRTR consists of measuring the degree to which an instrument yield reproducible score at different points in time assessed across a fixed and common time interval for all subjects. TRTR co-relations were based on the two-way mixed effect ICC coefficient estimated using the inter-rater reliability package, version 0.84.1. TRTR estimate of 0.7 and above indicated better retest reliability. TRTR was assessed among participants reporting no change on PGI-S between screening and baseline. PGI-S anchors are PRO specific, with a respiratory PGI-S (scale ranging from 1=not at all to 5=extremely severe, Higher scores=greater symptom severity) applied to the QOL-B respiratory domain (9-item scale ranging from 0 to 100, higher scores=fewer symptoms and better quality of life). As pre-specified in statistical analysis plan(SAP) for participants contributing to this outcome measure from INS-415 study,data were collected and analyzed for combined population in which ALIS and ELC groups were pooled.
Time Frame: From Screening to Baseline (Day -70 to Day 1)
Population: As pre-specified in the SAP, to adequately power the planned modern psychometric methods (MPMs) the cross-sectional validation sample was composed of a total of 97 participants enrolled in the INS-415 study (comprising of pooled ALIS + ELC data per planned analyses) who provided item-level QOL-B Respiratory domain data and Screening/Baseline data from the first 132 participants enrolled in the INS-416 study (NCT04677569) to yield a total sample of n=229.
Measure: Number; unit: ICC estimate
Groups:
- ALIS or ELC Along With Background Regimen (Azithromycin + Ethambutol): Combined Group: Participants received 590 mg of ALIS or ELC, a matching Placebo to ALIS, once daily. Participants also received the background regimen of azithromycin 250 mg and ethambutol 15 mg/kg tablets orally, once daily. Participants from both INS-415 and INS-416 were pooled for analysis in this combined group.
Arm/Group | ALIS or ELC Along With Background Regimen (Azithromycin + Ethambutol): Combined Group
Number analyzed (Participants) | 229
ICC estimate | 0.69

6. Primary Outcome: Assessment of TRTR Reported as the ICC Estimate Among Participants Reporting no Change on Fatigue PGI-S Score Applied to PROMIS F-SF 7a Score Between Screening and Baseline
Description: TRTR consists of measuring the degree to which an instrument yield reproducible score at different points in time assessed across a fixed and common time interval for all subjects. TRTR co-relations were based on the two-way mixed effect ICC coefficient estimated using the inter-rater reliability package, version 0.84.1. TRTR estimate of 0.7 and above indicated better retest reliability. TRTR was estimated using mean PROMIS F-SF 7a scores from participants who were stable as defined by a PGI-S-Fatigue change score of zero between screening and baseline. As pre-specified in the SAP, for participants contributing to this outcome measure from INS-415 study, data were collected and analyzed for combined population in which ALIS and ELC groups were pooled.
Time Frame: From Screening to Baseline (Day -70 to Day 1)
Population: As pre-specified in the SAP, to adequately power the planned MPMs the cross-sectional validation sample was composed of a total of 98 participants enrolled in the INS-415 study (comprising of pooled ALIS + ELC data per planned analyses) who provided item-level PROMIS F-SF 7a data and Screening/Baseline data from the first 132 participants enrolled in the INS-416 study to yield a total sample of n=230.
Measure: Number; unit: ICC estimate
Arm/Group | ALIS or ELC Along With Background Regimen (Azithromycin + Ethambutol): Combined Group
Number analyzed (Participants) | 230
ICC estimate | 0.76

7. Primary Outcome: Response Rate as Assessed by Within-Subject Meaningful Change (WSMC) for QOL-B Respiratory Symptoms Final Score Estimated Via Anchor-Based Methods and Validated Via Empirical Cumulative Distribution Functions (eCDFs)
Description: WSMC was estimated via change scores computed between Baseline and end of study (EOS) (Month 7). The estimated WSMC threshold of 14.81 points for the QOL-B Respiratory Symptom score (9-item scale ranging from 0 to 100, higher scores=fewer symptoms and better quality of life) as derived from anchor-based methods supplemented with eCDF curves was used for analysis. The percentage of participants and confidence intervals were estimated by standardized logistic regression with treatment group and history of mycobacterium avium complex (MAC) lung infection as factors in the model. Missing change from baseline at Month 7 was imputed by multiple imputation. The mean of all imputed values was used to derive response according to WSMC. Response rate was expressed in terms of percentage of participants and the percentages are rounded off to the nearest decimal.
Time Frame: Baseline to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
percentage of participants | 43.8 [29.8 to 57.8] | 33.3 [20.4 to 46.2]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.2819, Standardized Logistic Regression; Percentage Difference = 10.4, 95% CI 2-sided [-8.6 to 29.5] — The percentage difference and confidence intervals are estimated by standardized logistic regression with treatment group and history of MAC lung infection as factors in the model

8. Primary Outcome: Response Rate as Assessed by WSMC for PROMIS Fatigue Final Score Estimated Via Anchor-Based Methods and Validated Via eCDFs
Description: WSMC was estimated via change scores computed between Baseline and EOS (Month 7). The percentage of participants and confidence intervals were estimated by standardized logistic regression with treatment group and history of MAC lung infection as factors in the model. Missing change from baseline at Month 7 was imputed by multiple imputation. The mean of all imputed values was used to derive response according to WSMC. The estimated WSMC threshold of -4.00 points for the PROMIS Fatigue score as derived from anchor-based methods supplemented with eCDF curves was used for analysis. Response rate was expressed in terms of percentage of participants and the percentages are rounded off to the nearest decimal.
Time Frame: Baseline to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
percentage of participants | 35.5 [22.2 to 48.7] | 29.4 [17.1 to 41.6]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.5080, Standardized Logistic Regression; Percentage Difference = 6.1, 95% CI 2-sided [-11.9 to 24.1] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Percentage of Participants Achieving Culture Conversion by Month 6
Description: Culture conversion by Month 6 was defined as no MAC growth on agar media and broth media in all sputum cultures at 2 consecutive visits up to Month 6. Percentage of participants and confidence intervals were estimated by standardized logistic regression with treatment group and history of MAC lung infection as factors in the model. For the purpose of the estimation missing conversion status by Month 6 was imputed by multiple imputation. Percentages are rounded off to the nearest decimal.
Time Frame: Baseline to Month 6
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
percentage of participants | 80.6 [68.7 to 92.6] | 63.9 [50.2 to 77.6]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.0712, Standardized Logistic Regression; Percentage Difference = 16.7, 95% CI 2-sided [-1.4 to 34.9]

10. Secondary Outcome: Change From Baseline in QOL-B Respiratory Symptom Score at Month 7
Description: The QOL-B is a self-administered, PRO questionnaire used to assess symptoms, functioning, and health related quality of life in adults with lung conditions. The respiratory symptom domain of the QOL-B contains 9 items describing patient's self-assessment of her/his respiratory symptoms that affect daily life. For each of the 8 items (chest congestion, coughing, cough up mucus, shortness of breath with greater activity, wheezing, chest pain, shortness of breath when talking, woken up during night due to cough), scores ranged from 1 to 4 (1= lot, 2= moderate, 3= little, 4= not at all) and the sputum item based on the color ranged from 0=don't know,1=green with traces of blood/brownish dark,2=yellowish-green,3=clear to yellow,4=clear. The item scores were summed and then standardized on a 0 to 100-point scale to derive the domain score with higher scores representing fewer symptoms or better functioning and quality of life. Positive change from baseline indicates improvement.
Time Frame: Baseline to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
score on scale | 12.24 [7.96 to 16.53] | 7.76 [3.76 to 11.77]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.1073, ANCOVA; Least Square Mean Difference = 4.48, 95% CI 2-sided [-0.97 to 9.93]

11. Secondary Outcome: Change From Baseline in PROMIS F-SF 7a Score at Month 7
Description: as for outcome 4
Time Frame: Baseline to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
score on a scale | -2.1 [-3.4 to -0.8] | -1.6 [-2.9 to -0.3]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.6130, ANCOVA; Least Square Mean Difference = -0.4, 95% CI 2-sided [-2.2 to 1.3]

12. Secondary Outcome: Time to First Culture Conversion
Description: Time to first culture conversion was the number of months between first study drug intake and date of the first negative culture at or before Month 6 after adjustment for non-productivity. Participants without conversion at or before Month 6 are considered censored at the last visit with available culture assessment at or before Month 6.
Time Frame: Baseline to Month 6
Population: The ITT Analysis Set comprises all participants who were randomized. Overall number analyzed is the number of participants with culture conversion who had data available for analyses.
Measure: Median (Full Range); unit: months
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 39 | 40
months | 1.0 [1 to 5] | 2.0 [1 to 5]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.3542, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.79 to 1.92] — A Cox regression model was applied to calculate the hazard ratio. The model included effects for treatment and history of MAC lung infection (initial or subsequent)

13. Secondary Outcome: Time to First Negative Culture
Description: Time to first negative culture was the number of months from the date of first dose of study drug(s) to the date of first MAC culture negative post-baseline. Participants without negative culture were considered censored at the last visit with available culture assessment or at Month 7 whichever occurred first.
Time Frame: Baseline to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized. Overall number analyzed is the number of participants with a negative culture.
Measure: Median (Full Range); unit: months
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 45 | 44
months | 1.0 [1 to 3] | 1.0 [1 to 7]
Statistical Analysis 1: Comparison: ALIS + Background Regimen (Azithromycin + Ethambutol) vs ELC + Background Regimen (Azithromycin + Ethambutol); Test type: Superiority; p = 0.1583, Regression, Cox; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.89 to 2.06] — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Percentage of Participants Who Develop a MAC Isolate With Amikacin Minimum Inhibitory Concentration (MIC) ≥ 128 Micrograms Per Millliliter (µg/mL) at More Than 1 Visit
Time Frame: Up to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
percentage of participants | 0 | 0

15. Secondary Outcome: Recurrence of MAC (Relapse) Assessed as Percentage of Participants Who Achieved Culture Conversion With a Subsequent at Least One MAC Positive Culture in Agar Media or Broth Media in at Least 2 Consecutive Visits
Description: Culture conversion for this outcome measure was defined as MAC culture negative at 2 consecutive visits before or at Month 5 during the treatment period. The positive culture was defined as at least 1 MAC positive culture in agar media or positive cultures in broth media in at least 2 consecutive visits. Percentages are rounded off to the nearest decimal.
Time Frame: Baseline to Month 7
Population: The ITT Analysis Set comprises all participants who were randomized. Overall number analyzed is the number of participants who had conversion before or at Month 5 with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 39 | 40
percentage of participants | 5.1 | 22.5

16. Secondary Outcome: Recurrence of MAC (New Infection) Assessed as Percentage of Participants Who Achieved Culture Conversion With a Subsequent at Least One MAC Positive Culture in Agar Media or Broth Media in at Least 2 Consecutive Visits
Description: as for outcome 15
Time Frame: Baseline to Month 7
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 39 | 40
percentage of participants | 5.1 | 25.0

17. Secondary Outcome: Number of Participants Who Experience Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs are AEs that occurred on or after the date of first dose of study drugs and within 28 days after the end of treatment.
Time Frame: Baseline to Month 7
Population: The Safety Analysis Set comprises all participants who were randomized and received at least 1 dose of ALIS, ELC, azithromycin or ethambutol.
Measure: Count of Participants; unit: Participants
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
Number analyzed (Participants) | 48 | 51
Participants | 44 | 41

ADVERSE EVENTS:
Time Frame: Baseline to Month 7
Description: The Safety Analysis Set comprises all participants who were randomized and received at least 1 dose of ALIS, ELC, azithromycin or ethambutol.
Arm/Group | ALIS + Background Regimen (Azithromycin + Ethambutol) | ELC + Background Regimen (Azithromycin + Ethambutol)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 7/48 | 3/51
Other Adverse Events (participants affected / at risk) | 38/48 | 33/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALIS + Background Regimen (Azithromycin + Ethambutol) (N=48) | ELC + Background Regimen (Azithromycin + Ethambutol) (N=51)
Bronchiolitis (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALIS + Background Regimen (Azithromycin + Ethambutol) (N=48) | ELC + Background Regimen (Azithromycin + Ethambutol) (N=51)
Tinnitus (Ear and labyrinth disorders) | 2 | 4
Vision blurred (Eye disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 13 | 13
Nausea (Gastrointestinal disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 5 | 6
Asthenia (General disorders) | 2 | 5
COVID-19 (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3
Weight decreased (Investigations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 5 | 6
Dizziness (Nervous system disorders) | 2 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 20 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT04677543/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT04677543/SAP_001.pdf